CLINICAL TRIAL: NCT00934011
Title: Comparative Study of C-reactive Protein vs. Procalcitonin to Guide Antibiotic Therapy in Patients With Severe Sepsis and Septic Shock Admitted to the Intensive Care Unit.
Brief Title: Use of Inflammatory Biomarkers to Guide Antibiotic Therapy in Patients With Severe Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other)
Responsible Party: Principal Investigator, Vandack Alencar Nobre, Associate Professor, PhD, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO_Protocol01
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2012-06

CONDITIONS: Severe Sepsis; Septic Shock
Keywords: C-reactive protein; procalcitonin; sepsis; antibiotic therapy
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 - C-reactive protein (CRP) guided ab therapy (Experimental): Intervention on antibiotic therapy will be based on circulating CRP levels
  Interventions: Other: C-reactive protein guided antibiotic therapy
- Group 2 - procalcitonin (PCT) guided ab therapy (Active Comparator): Intervention on antibiotic therapy will be based on circulating PCT levels
  Interventions: Other: Procalcitonin guided antibiotic therapy

INTERVENTIONS:
Other: C-reactive protein guided antibiotic therapy — plasma CRP measurement to guide the duration of antibiotic therapy
  Arms: Group 1 - C-reactive protein (CRP) guided ab therapy
Other: Procalcitonin guided antibiotic therapy — plasma PCT measurement to guide the duration of antibiotic therapy
  Arms: Group 2 - procalcitonin (PCT) guided ab therapy

SUMMARY:
In this study the investigators aim to test if C-reactive protein (CRP)or procalcitonin(PCT) - guided strategy allows to reduce the antibiotic use in patients wiht severe sepsis and septic shock. Therefore, the safety of this intervention will be carefully measured.

DETAILED DESCRIPTION:
Methods

* Patients and settings: Prospective controlled randomized open interventional study of antibiotic therapy in adult with severe sepsis or septic shock, admitted to the intensive care unit.

The study will be conducted in the intensive care unit (ICU) of the University Hospital Risoleta Tolentino Neves of the Federal University of Minas Gerais, Brazil. This is a 30-bed ICU with medical and surgical patients. All patients with suspected severe sepsis or septic shock admitted to the ICU will be assessed for eligibility. Patients developing severe sepsis or septic shock during their ICU stay will be also considered for enrollment.

Cultures of urine, blood, bronchoalveolar lavage ﬂuid, and tracheal aspirates will be performed on admission and during ICU stay as clinically indicated. Blood gases and imaging exams will also be performed as clinically indicated, similarly in both groups.

* Interventions:

All adult (> 17 years old) patients with diagnosis of severe sepsis or septic shock will receive initial antibiotic therapy based on local guidelines and susceptibility patterns, according to the decision of the treating physician. They will have circulating PCT and CRP levels measured at baseline and daily until day 4 in both groups.

Eligible patients will be reassessed on day 4 and randomized at 1:1 basis to one of the two groups since any exclusion criteria (see below) is present at that time:

Group 1 - CRP group: the duration of antibiotic therapy will be based on circulating CRP levels.

Group 2 - PCT group: the duration of antibiotic therapy will be based on circulating PCT levels.

Patients enrolled in the study will undergo daily measurements of plasma CRP (Dry Chemistry - Johnsons & Johnsons) and PCT (BRAHMS PCT VIDAS) levels up to stopping antibiotic therapy, every 48hr for two measurements in patients remaining in the ICU, and then, every 5 days.Patients will be followed up 28 days, or until death or hospital transference, which comes first. PCT and CRP results will be released in sealed envelopes. During the study period, only the results corresponding to the patient randomization group will be open; i.e., CRP for CRP group patients and PCT for PCT group patients.

- Criteria for antibiotic interruption:

The investigators will propose the interruption of antibiotics if:

1. The patients is clinically stable, without signs of active infection
2. CRP group: a relative reduction of 50% in baseline CRP levels, or a value lower than 25mg/dl is reached.
3. PCT group: a relative reduction of 90% in baseline PCT levels, or if a absolute value lower than 0.1 ng/ml is reached.

The final decision regarding antibiotic therapy will be always let to the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* age > 17 years
* patients in intensive care unit
* signed informed consent
* suspected or confirmed severe sepsis or septic shock

Exclusion Criteria:

* Infections caused by Listeria spp, Legionella pneumophilia, Mycobacterium tuberculosis
* Bacteremia due S. aureus
* Infections requiring prolonged therapies, such as endocarditis, cerebral abscess, chronic osteomyelitis
* Suspected or confirmed infection caused by virus, parasites
* Infections caused by P. aeruginosa ou A. baumannii
* Severe immunosuppression (ex: AIDS, post bone-marrow transplant,cystic fibrosis)
* Traumatism latest five days
* Surgery latest 5 days
* Carcinoid tumor, lung cancer, medullary thyroid cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2009-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Duration of antibiotic therapy for the first episode of infection | 28 days
Total antibiotic exposure days per 1,000 days | 28 days
Days alive without antibiotics | 28 days

SECONDARY OUTCOMES:
All cause 28-day mortality | 28 days
clinical cure rate | 28 days
Infection relapse (diagnosed less than 48h after antibiotic discontinuation) | 48 hours
Length of ICU stay | Whole hospitalization
Nosocomial infection rate | 28 days
In-hospital mortality | 28 days
sepsis-associated death | 28 days
Nosocomial superinfection (diagnosed more than 48hous after discontinuation of the antibiotic therapy given to the first episode of infection) | 28 days
Isolation of resistant bacteria | 28 days
Length of hospital stay | The whole hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Vandack A Nobre, PhD, Principal Investigator — Medical School of the Federal University of Minas Gerais; Carolina F Oliveira, MD, Study Chair — Idem; Fernando A Botoni, PhD, Study Chair — Idem
Locations (1):
- Hospital das Clínicas - Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Results published in the Critical Care Medicine, 2013

REFERENCES:
- [Derived] Oliveira CF, Botoni FA, Oliveira CR, Silva CB, Pereira HA, Serufo JC, Nobre V. Procalcitonin versus C-reactive protein for guiding antibiotic therapy in sepsis: a randomized trial. Crit Care Med. 2013 Oct;41(10):2336-43. doi: 10.1097/CCM.0b013e31828e969f. PMID 23921272